CLINICAL TRIAL: NCT06089317
Title: Traditional Chinese Medicine Ultrasonic Atomization Treatment for Dry Eye Disease: A Randomized, Double-masked, Placebo-controlled Trial
Brief Title: Traditional Chinese Medicine Ultrasonic Atomization Treatment for Dry Eye Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Kelvin Kam-lung Chong, MD, Associate Professor, Department of Ophthalmology and Visual Sciences, CUHK, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMDF-21B2005A_R1
Record Dates: First submitted 2023-10-13; First posted 2023-10-18 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Dry Eye Syndromes
Keywords: Dry Eye Syndromes; Traditional Chinese Medicine; Ultrasonic Atomization; Randomized Controlled Trial
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Lubricant Eye Drops

STUDY DESIGN:
Intervention Model Description: A total of 200 subjects with mild to moderate DED will be recruited. Only one eye of recruited subjects with the shorter NIBUT will be selected and analyzed as the study eye. The subjects will be randomly divided into TCM compound decoction (CD) group, dendrobium caulis (DC) group, houttuynia cordata (HC) group, placebo atomization (PA) group, and artificial tears (AT) group equally. An online-based clinical trial randomization tool with a permuted block and stratification randomization method is applied for the randomization, and block sizes are randomly chosen. Stratification variances is sex and age.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Compound Decoction (CD) group (Active Comparator)
  Interventions: Drug: TCM ultrasonic atomization treatment with herbal Compound Decoction (CD); Drug: Artificial Tears (AT)
- Dendrobii Caulis (DC) group (Active Comparator)
  Interventions: Drug: TCM ultrasonic atomization treatment with Dendrobii Caulis (DC); Drug: Artificial Tears (AT)
- Houttuynia Cordata (HC) group (Active Comparator)
  Interventions: Drug: TCM ultrasonic atomization treatment with Houttuynia Cordata (HC); Drug: Artificial Tears (AT)
- Placebo Atomization (PA) group (Placebo Comparator)
  Interventions: Drug: Placebo TCM ultrasonic atomization treatment (PA); Drug: Artificial Tears (AT)
- Artificial Tears (AT) group (Other)
  Interventions: Drug: Artificial Tears (AT)

INTERVENTIONS:
Drug: TCM ultrasonic atomization treatment with herbal Compound Decoction (CD) — The subjects will receive TCM ultrasonic atomization treatment with the ultrasonic nebulizer (WH-2000, YueHua, China) 6 days a week, once daily, 10 minutes per session, for 4 weeks. The solution for atomization of the CD group is TCM compound decoction.
  The prescription of atomization solution in the CD group contains Honeysuckle flower (金銀花) 5g, Chrysanthemum flower (菊花) 5g, Pale betterflybush flower (密蒙花) 5g, Mild mint herb (薄荷) 5g, Barbary wolfberry fruit (枸杞子) 10g, and Ophiopogon japonicus (麥冬) 5g.
  Subjects will be treated with hypromellose 0.3% w/v eye drops four times per day too.
  Arms: Compound Decoction (CD) group
Drug: TCM ultrasonic atomization treatment with Dendrobii Caulis (DC) — The subjects will receive TCM ultrasonic atomization treatment with the ultrasonic nebulizer (WH-2000, YueHua, China) 6 days a week, once daily, 10 minutes per session, for 4 weeks. The solution for atomization of the DC group is Dendrobii Caulis extracts.
  The prescription of the DC group contains Dendrobium (石斛) 35g.
  Subjects will be treated with hypromellose 0.3% w/v eye drops four times per day too.
  Arms: Dendrobii Caulis (DC) group
Drug: TCM ultrasonic atomization treatment with Houttuynia Cordata (HC) — The subjects will receive TCM ultrasonic atomization treatment with the ultrasonic nebulizer (WH-2000, YueHua, China) 6 days a week, once daily, 10 minutes per session, for 4 weeks. The solution for atomization of the HC group is Heartleaf Houttuynia Herb extracts.
  The prescription of the HC group contains Heartleaf Houttuynia Herb(魚腥草) 35g.
  Subjects will be treated with hypromellose 0.3% w/v eye drops four times per day too.
  Arms: Houttuynia Cordata (HC) group
Drug: Placebo TCM ultrasonic atomization treatment (PA) — The subjects will receive TCM ultrasonic atomization treatment with the ultrasonic nebulizer (WH-2000, YueHua, China) 6 days a week, once daily, 10 minutes per session, for 4 weeks. The solution for atomization of the PA group is low-concentration compound decoction (5%) same with the CD group.
  Subjects will be treated with hypromellose 0.3% w/v eye drops four times per day too.
  Arms: Placebo Atomization (PA) group
Drug: Artificial Tears (AT) — The subjects will receive lubricant eye drop (Hypromellose 0.3% w/v Eye Drops) four times per day only.

SUMMARY:
Dry eye disease (DED) is the most prevalent ocular surface disease worldwide. Standard treatments like artificial tears show limited effect. Regarding the ultrasonic atomization, the ultrasonic nebulizer produces consistent steam from the solution with a treatment effect delivered to the ocular surface. We aim to evaluate the effectiveness and safety of traditional Chinese medicine (TCM) ultrasonic atomization as an adjuvant treatment for DED.

This is a randomized double-masked, active- and placebo-controlled trial. 200 subjects will be equally assigned to the herbal compound decoction(CD) group, dendrobium caulis (DC) group, houttuynia cordata (HC) group, placebo atomization(PA) group, and artificial tear (AT) group by stratified permuted block randomization.

Subjects of CD, DC, HC, and PA groups will receive TCM ultrasonic atomization treatment (6 times/week). All patients will receive hypromellose 0.3% w/v lubricant eye drops for a 1-week wash-out and a 4-month follow-up period. Outcomes included non-invasive tear break-up times, corneal and conjunctival fluorescein staining, and other dry eye-related parameter examined by LipiView II Ocular Surface Interferometer, OCULUS® Keratograph 5M, and slit lamp biomicroscope evaluated by masked clinical assessors at baseline, week 1, 2, 3, 4 and month 2, 3, 4. The other subjective questionnaires like the Ocular Surface Disease Index (OSDI) questionnaire are also selected.

ELIGIBILITY:
Inclusion criteria:

1. At least one eye of subjects meets DED diagnostic criteria as the Tear Film and Ocular Surface Society (TFOS) Dry Eye Workshop (DEWS II); and
2. Ocular Surface Disease Index (OSDI)≥13 and <33; and
3. The age range between years 18-80, no sex limitation; and
4. Symptoms of dry eye for at least 6 months; and
5. Can complete the questionnaires independently and understand Chinese or English.

Exclusion criteria:

1. Had or currently suffering from other concomitant ocular surface diseases, including chronic conjunctivitis, ocular rosacea, cicatricial pemphigoid, graft-versus-host disease, limbal stem cell deficiency, and severe ocular allergy;
2. Received any refractive surgery and corneal surgery before, including corneal transplant; or any eye surgery in the past 6 months;
3. Receiving DED-related medications, including topical steroid eyedrops, topical antibiotics, topical cyclosporin A, and topical diquafosol;
4. Received intense pulsed laser (IPL) or vectored thermal pulsation (VTP) therapy in the past 12 months;
5. Received topical antiglaucomatous treatment in the past 12 months
6. Plans to use contact lenses during treatment and follow-up periods or used contact lenses 2 weeks before the baseline measurement and recruitment;
7. Had or currently suffering from severe cardiopulmonary disease, liver and kidney dysfunction, and severe blood system diseases;
8. Suffering from glucose-6-phosphate dehydrogenase deficiency (G6PD);
9. Had or currently suffering from specific respiratory diseases, e.g. emphysema, bronchitis, asthma, chronic obstructive pulmonary disease, bronchial dilatation;
10. Has adverse reaction history to herbs used in this study before;
11. Whose TCM constitution is manifested as "yang-deficiency" or diagnosed by TCM practitioners that their TCM syndrome is not suitable for the atomization treatment;
12. Pregnancy, preparation for pregnancy, or lactation;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-07-28 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in the Ocular Surface Disease Index (OSDI) | baseline to 4th week
  The Ocular Surface Disease Index (OSDI) is a 12-item symptom frequency-based questionnaire. It is self-administered to assess DED-related symptoms and severity.
  The final OSDI score is calculated by dividing the product of the total sum of the score and 25 by the total number of answered questions, with a range from 0 to 100. The score reflects the severity of DED(normal: 0-12, mild: 13-22, moderate: 23-32, severe: >33).
Change in Non-invasive Tear Break-up Times (NIBUT) | baseline to 4th week
  The non-invasive tear break-up time (NIBUT) will be measured by the OCULUS Keratograph® 5M (Oculus, Wetzlar, Germany). Subjects will be instructed to keep their eyes on as much as possible during the examination. First and average NIBUT will be recorded by the machine accordingly.
  Shortening NIBUT(< 10 seconds) suggests instability of the tear film.

SECONDARY OUTCOMES:
Change in Ocular Surface Disease Index (OSDI) | 4 months
  The Ocular Surface Disease Index (OSDI) is a 12-item symptom frequency-based questionnaire. It is self-administered to assess DED-related symptoms and severity.
  The final OSDI score is calculated by dividing the product of the total sum of the score and 25 by the total number of answered questions, with a range from 0 to 100. The score reflects the severity of DED: normal: 0-12, mild: 13-22, moderate: 23-32, severe: >33).
Change in symptom Assessment iN Dry Eye (SANDE, modified) | 4 months
  Symptom Assessment iN Dry Eye (SANDE) questionnaire is a 2-item frequency- and severity-based visual analog scale. It is self-administered to evaluate the frequency and severity of dry eye symptoms.
  The final SANDE score is calculated by obtaining the square root of the product of the frequency of symptoms score and the severity of symptoms score, with a range from 0 (minimal degree of dry eye symptoms) to 100 (maximal degree of dry eye symptoms)
Change in 36-Item Short Form Health Survey (SF-36) | 4 months
  The 36-Item Short Form Health Survey (SF-36) is a 36-item self-administered questionnaire, with 8 domains included: physical functioning (PF), role physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MH). The physical health sub-scale and Mental health sub-scale will be graded respectively.
Change in the Work Productivity and Activity Impairment Questionnaire: General Health V2.0 (WPAI:GH) | 4 months
  The Work Productivity and Activity Impairment Questionnaire: General Health V2.0 (WPAI: GH) is a 6-item questionnaire that measures impairments in work and activities.
Change in Non-Invasive Tear Break Up Times (NIBUT) | 4 months
  Non-Invasive tear break up time (NIBUT) will be measured by the OCULUS Keratograph® 5M (Oculus, Wetzlar, Germany) in both eyes. Participants were instructed to keep their eyes on as much as possible during the examination. First and average NIKBUTs will be recorded by the machine.
  Shortening NIBUT(< 10 seconds) suggests instability of the tear film.
Changes in Tear Meniscus Height (TMH) | 4 months
  The tear meniscus height (TMH) will be measured by the OCULUS Keratograph® 5M (Oculus, Wetzlar, Germany).
Changes in Bulbar Redness | 4 months
  Bulbar conjunctival hyperaemia is automatically evaluated the Keratograph 5M (OCULUS, Wetzlar, Germany) according to the JENVIS grading scale from 0 to 4.
Changes in Lipid Layer Thickness | 4 months
  The lipid layer thickness (LLT) of the tear film will be determined with the LipiView ® II Ocular Surface Interferometer (TearScience, Morrisville, NC). Minimum, Maximum, and Average thickness in nanometers (nm) will be measured.
Changes in Partial Blinking Rate | 4 months
  The partial blinking rate will be reported as the percentage of incomplete blinks. The total and partial blinking times will be automatically recorded by the LipiView ® II Ocular Surface Interferometer (TearScience, Morrisville, NC).
Changes in Meiboscore | 4 months
  The meiboscore grading will be based on the infrared meibography captured by the LipiView ® II Ocular Surface Interferometer (TearScience, Morrisville, NC). Both superior and inferior eyelids will be recorded. The result will be graded by a masked assessor.
  The grading scheme is a 3-point scale (grade 0, no meibomian gland atrophy; grade 1, less than 1/3 area of glands lost; grade 2, 1/3-2/3 area of glands lost; grade 3, more than 2/3 area of glands lost)
Change in Tear Film Breakup Time (TBUT) | 4 months
  The tear film breakup time (TBUT) is the time of the initial breakup of the tear film after a full blink. 2% Sodium fluorescein will be instilled in both eyes of the subjects. A masked follow-up assessor will do the examination via the slit lamp with a blue cobalt light. The TBUT will be measured three times with a stopwatch and taken on average.
Change in Corneal and Conjunctival Fluorescein Staining | 4 months
  Fluorescein sodium liquid will be instilled on the ocular surface. After 3 minutes, the corneal and conjunctival punctate epithelial erosions will be observed and graded via the slit lamp biomicroscope with a blue cobalt light.
  The Oxford Grading System is selected for grading. The severity will be divided into 6 grades (Grade 0, absent; Grade 1, minimal; Grade 2, mild; Grade 3, moderate; Grade 4, marked; Grade 5, severe)
Change in Expressibility of Meibomian Glands in the Meibomian Glands Yielding Liquid Secretion (MGYLS) (the inferior eyelid) | 4 months
  Expressibility of the inferior eyelid meibomian glands is assessed with the Meibomian Gland Evaluator (TearScience, North Carolina, USA) applied inferior to central aspects of the inferior eyelid margin. The result is graded by a masked assessor.
  The meibomian glands yielding liquid secretion (MGYLS) is the total number of glands that yield lipid secretions at the central aspects of the eyelid margin.
Change in Quality of Expressed Meibum | 4 months
  The meibomian gland evaluator will be applied to the central aspects of the inferior eyelid margin. The result will be graded by a masked assessor.
  Each gland in each area will be assessed for expressibility and graded according to a 4-point scale: grade 0, no secretion; grade 1, inspissated/ toothpaste-like expression; grade 2, cloudy fluid secretion; and grade 3, clear fluid/normal secretion. The sum scores of 5 glands will be between 0 and 15.
Change in Lid Margin and Eyelash Abnormalities | 4 months
  Lid margin and eyelash abnormalities will be accessed by a slit lamp, including telangiectasia, meibomian gland capping, Demodex lash cylindrical collarettes, staphylococcal lash crusting, and seborrheic lash crusting.
  All items will be graded based on a four-point scale: grade 0, absent; grade 1, mild; grade 2, moderate; grade 3, severe.
Change in Tear Film Osmolarity (TFO) | 4 months
  The tear film osmolarity (TFO) is measured by the ScoutPro™ Osmolarity System (TearLab , San Diego, CA) via the disposable test card in both eyes.
  The normal osmolarity was considered as lower than 308 mOsm/L in both eyes. A difference more than 8 mOsm/L between two eyes reflects the stability of the tear film.
Changes in Schirmer I test | 4 months
  The Schirmer I test (ST) will be performed by sterile standard filter paper strips without anesthesia. The filter paper strips will be gently put on the temporal side of both lower eyelids for 5 minutes. The wetting length by tears in each strip will be recorded in nanometers (mm) by a masked assessor.
  The strips will be collected in sterile centrifuge tubes respectively for further laboratory tests.
Changes in Matrix metallopeptidase 9 (MMP-9) | 4 months
  The MMP-9 enzyme-linked immunosorbent assay (ELISA) development kit (Invitrogen, Carlsbad, CA)) will be applied for measurement of the concentration of MMP-9 in participants' tears.
Adverse events (AEs) | 4 months
  The adverse events (AEs) will be the number of incidents based on a checklist of symptoms, signs, and diseases by patients' reporting, slit-lamp examination, or doctor's diagnosis.

OTHER OUTCOMES:
Intraocular Pressure (IOP) | 4 months
  The intraocular pressure of the eyes will be assessed by a non-contact tonometer.
Best Corrected Visual Acuity (BCVA) | 4 months
  Best corrected visual acuity (BCVA) is examined by a standard visual acuity chart.
Change in Posterior Subcapsular of Lens | 4 months
  The Lens Opacities Classification Systems (LOCS III) will be applied for lens grading.
  The posterior subcapsular (P) cataract will be graded referring to five retroillumination images: P1-P5.
Change in Nuclear Color (NC) of Lens | 4 months
  The Lens Opacities Classification Systems (LOCS III) will be applied for lens grading.
  Nuclear color (NC) will be graded referring to referring to six slit-lamp images: NC1-NC6.
Change in Cortical Cataract (C) of Lens | 4 months
  The Lens Opacities Classification Systems (LOCS III) will be applied for lens grading.
  Cortical cataract (C) will be graded referring to five retroillumination images: C1-C5.
Change in Nuclear Opalescence (NO) of Lens | 4 months
  The Lens Opacities Classification Systems (LOCS III) will be applied for lens grading.
  Nuclear opalescence (NO) will be graded referring to six slit-lamp images: NO01-NO06.
Change in Central Corneal Thickness (CCT) of Corneal Endothelium | 4 months
  Central corneal thickness will be measured with a non-contact specular microscope (Nidek CEM-530, NIDEK Co., Ltd. Japan).
Change in Corneal Endothelial Cell Density (CD) of Corneal Endothelium | 4 months
  Corneal endothelial cell density will be measured with a non-contact specular microscope (Nidek CEM-530, NIDEK Co., Ltd. Japan).
Change in Number of Cells Counted (NUM) of Corneal Endothelium | 4 months
  Number of cells counted will be measured with a non-contact specular microscope (Nidek CEM-530, NIDEK Co., Ltd. Japan).
Constitution in Chinese Medicine Questionnaire (CCMQ) | -1 week
  Constitution in Chinese Medicine Questionnaire (CCMQ) is a self-administered questionnaire with 60 items. It will be applied to classify a person's traditional Chinese medicine constitution out of 9 pre-defined types.
Change of α-diversity in Ocular Surface Microbiome | 4 months
  Each eye will be sampled by a sterile, polyester swab on the inferior fornix of the conjunctiva. The swabs will be placed in 2 mL microcentrifuge tubes at 4 °C. Extraction will be performed by laboratory staff, then the sample will be transferred to -80 °C laboratory freezer for long-term storage before further gene expression tests. After genomic DNA extraction from conjunctival swab samples for 16S rRNA sequencing, the resulting amplicons will be filtered, clustered into operational taxonomic units (OTUs) and taxonomically classified using reference databases. The α-diversity will be calculated and reported as ordination plots.
Change of β-diversity in Ocular Surface Microbiome | 4 months
  Each eye will be sampled by a sterile, polyester swab on the inferior fornix of the conjunctiva. The swabs will be placed in 2 mL microcentrifuge tubes at 4 °C. Extraction will be performed by laboratory staff, then the sample will be transferred to -80 °C laboratory freezer for long-term storage before further gene expression tests. After genomic DNA extraction from conjunctival swab samples for 16S rRNA sequencing, the resulting amplicons will be filtered, clustered into operational taxonomic units (OTUs) and taxonomically classified using reference databases. The β-diversity will be calculated and reported as ordination plots.
Relative Abundance in Ocular Surface Microbiome | 4 months
  Each eye will be sampled by a sterile, polyester swab on the inferior fornix of the conjunctiva. The swabs will be placed in 2 mL microcentrifuge tubes at 4 °C. Extraction will be performed by laboratory staff, then the sample will be transferred to -80 °C laboratory freezer for long-term storage before further gene expression tests. After genomic DNA extraction from conjunctival swab samples for 16S rRNA sequencing, the resulting amplicons will be filtered, clustered into operational taxonomic units (OTUs) and taxonomically classified using reference databases. The relative abundance will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Kelvin KL Chong, MBChB, Principal Investigator — Chinese University of Hong Kong
Locations (4):
- Hong Kong (4):
  - The Chinese University of Hong Kong Eye Centre (CUHKEC), Kowloon
  - Hong Kong Eye Hospital, Kowloon
  - The CUHK Medical Centre (CUHKMC), Shatin
  - Prince of Wales Hospital, Shatin